CLINICAL TRIAL: NCT01816100
Title: The Effect of Exercise on Strength and Mobility and Corresponding CNS Plasticity in Multiple Sclerosis Patients: A Multimodal Neuroimaging Investigation
Brief Title: The Effect of Exercise on Strength and Mobility and Corresponding CNS Plasticity in Multiple Sclerosis Patients
Acronym: remapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0039-13-EP
Record Dates: First submitted 2013-02-25; First posted 2013-03-21 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; exercise; MEG; DTI; Brain changes
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise session (Experimental): 6 months weight resistance session, with before/after evaluations by MEG and DTI. Fifty minute exercise sessions, twice weekly will be done. Each session will rotate between 3 separate exercise protocols: Static weights, free weights and balance. Exercises will be done with each extremity independently. For consistency and convenience, the resistance training will be performed at Fast Forward Gym, Omaha, NE.
  The primary outcome exercise data include strength and endurance
  Interventions: Other: specifically design 6 month resistance training program; Behavioral: 6 months weight resistance and balance program

INTERVENTIONS:
Other: specifically design 6 month resistance training program — Data will be kept on the number of repetitions and amount of weight per exercise session See intervention description
  Other Names: 6 months weight resistance session,
Behavioral: 6 months weight resistance and balance program — 3 phases first phase-strength improvement using stationary machines second phase-time is divided between stationary machines, balance, dexterity third phase-free weight movements
  Other Names: 50-minute, biweekly sessions for 6 months

SUMMARY:
This study is a unique blend of new technologies never used in combination with individuals diagnosed with Multiple Sclerosis (MS). The results of this research will define changes in brain activity, functional brain activation and diffusion in the brain following 6 months of structured weight resistance and balance training. Positive changes would indicate that the therapy has ignited brain plasticity and may drive the brain to repair itself. These changes to the brain may affect recovery as a result of neuroplasticity, neuroprotection, and slowing of neural degeneration. No other trials have been published evaluating brain plasticity utilizing diffusion tensor imaging (DTI) and magnetoencephalography (MEG) in subjects with MS undergoing physical training. DTI has demonstrated the ability to find changes (plasticity) that occur in the brain and using the MEG findings to focus the DTI analysis will optimize the capacity to detect changes secondary to therapy. This quantification will give a better understanding of the repair that goes on in the brain, and may potentially revolutionize the field of the central nervous system (CNS) rehabilitation. One of the most innovative aspects of this study is the full integration of clinical neurobehavioral metrics and functional imaging data in conjunction with a proven MS therapy along with quality of life indicators. This approach will allow new links to be illuminated as the trajectories of functional and structural brain changes (neuroplasticity) are meshed with clinical improvement indices collected visit-by-visit. This study will also compare disease modifying treatments (DMTs) and their effect(s) on indices of brain plasticity and cognitive and behavioral assessments.

DETAILED DESCRIPTION:
Rationale MEG is a direct measure of ongoing neurophysiological activity and is appropriate because of spatiotemporal resolution of measurements and immunity of the technique to vascular biases that contaminate functional MRI imaging of MS patients.4 MEG will help to illuminate the brain bases of motor deficits that exist relative to healthy controls and show how the improvements observed behaviorally are reflected in the brain activity that underlies those improvements. Since DTI has demonstrated the ability to find changes (plasticity) that occur in the brain in patients, it is very promising that DTI will be able to detect evidence of neuroplasticity in our research population.5 Using the MEG findings to sharpen the DTI analysis, a very powerful combination, will optimize the ability to detect and understand changes.

Objectives Specific Aim 1 - Determine if there are activation differences (see below) in the neural regions serving motor function during basic movements using MEG in a group of MS patients, comparing MS affected portions of the brain versus non-affected.

Specific Aim 2 - Determine the effect of a specific 6 month resistance and balance exercise program on activation in sensorimotor brain areas using MEG, and correlate changes in these neural indices with those of specific movement and balance.

Specific Aim 3 - Determine the effect of a specific 6 month resistance and balance exercise program on brain diffusivity and fractional anisotropy using DTI and correlate changes in these metrics with improvement in strength and balance measures in subjects with MS, comparing MS affected portions of the brain versus non-affected areas..

Specific Aim 4 - Determine whether increased fiber integrity (fractional anisotropy) along the corticospinal tract is reflected in MEG activation metrics of the primary motor cortex from baseline to 6 months in subjects with MS enrolled in the three-month resistance and balance exercise program.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of relapsing/remitting or secondary progressive MS by McDonald Criteria (for patient groups)
* Competent to give informed consent.
* ≥ 19 years and <65 years of age.
* EDSS score <7.0 and able to walk 25 feet with or without a cane.
* Willingness to comply with the evaluation schedule for the study. This includes participation in a bi-weekly standardized structured resistance training and separate data collections done at each time point (baseline and 3 months).
* Evidence that the MS patient's physical and neurological examinations are "clinically acceptable." Clinically acceptable is defined as those clinical findings or conditions that would not place the patient in undue risk by participating and which would not interfere with outcome measures of the study.

Exclusion Criteria:

* Unable to give informed consent.
* Unable or unwilling to sign safety waiver.
* EDSS score ≥7 or are unable to walk 25 feet with the use of a cane
* Unwilling or unable to complete the exercise program and other aspects of the study (e.g., not keeping appointments, lack of active participation in the exercise sessions, or displaying inability to follow instructions allowing appropriate exercise advancement).
* Pregnant, breastfeeding or within 3 months post partum at initiation of study.
* Have any other disability that would affect balance and/or mobility.
* Have any other neurological or neurodegenerative disorders.
* Have any other conditions, clinical findings or reason that deems the subject unsuitable for enrollment into the study.
* Have an implantable device or history of metal in body.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Determine activation differences in neural regions serving motor function | measure after 6 months training session
  Determine activation differences in the neural regions serving motor function using MEG in a group of MS patients, comparing MS affected portions of the brain versus non-affected .Comparison of MEG and DTI measures and whether changes occur after an exercise intervention.

SECONDARY OUTCOMES:
Effect of a 6 month resistance and balance program on activation in sensorimotor brain areas | following 6 months of exercise sessions
  Determine effect of a 6 month resistance and balance program on activation in sensorimotor brain areas using MEG, and correlate changes in these neural indices with those of specific movement and balance.

OTHER OUTCOMES:
Effect of a 6 month resistance and balance program on brain diffusivity and fractional anisotropy | Following 6 month exercise session
  Determine effect of a 6 month resistance and balance program on brain diffusivity and fractional anisotropy using DTI and correlate changes with improvement in strength and balance measures in subjects with MS.

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Filipi, PhD, APRN, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States